CLINICAL TRIAL: NCT05942937
Title: National Prisons Hepatitis Education Project: Research Evaluation
Acronym: HepPEd
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Australasian Society for HIV Viral Hepatitis and Sexual Health Medicine (ASHM) (Unknown); Justice health, corrections, and hepatitis and drug-user organisations in each Australian state and territory (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VISP2101
Record Dates: First submitted 2023-04-21; First posted 2023-07-12 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: HCV
Keywords: Hepatitis C; Public Health; Health Service; Prison; Education
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: This is a single group, non-randomised, before-and-after trial of an education intervention being conducted in three to six selected prisons in Australia.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole-of-prison education intervention (Experimental): The HepPEd Program will saturate the entire prison during a 3-month intervention phase.
  Interventions: Other: Education Intervention (The HepPEd Program)

INTERVENTIONS:
Other: Education Intervention (The HepPEd Program) — All healthcare providers, correctional officers, and people in prison (HepPEd Program target audience groups) at each participating site are anticipated to be exposed to the HepPEd Program over the course of the three-month education intervention phase.
  The HepPEd Program involves a suite of multi-modal resources targeting each target audience group and a peer education program (for correctional officer and people in prison groups only). The HepPEd Program resources will be delivered in an informal, mass education-style, as well as in peer to peer format.

SUMMARY:
The National Prisons Hepatitis Education Program (HepPEd Program) is a national, prison-based hepatitis C health literacy education program for healthcare providers, correctional officers, and people in prison. The HepPEd Program aims to improve the public health literacy of the prison sector regarding hepatitis C in prisons.

The HepPEd: Research Evaluation aims to evaluate the impact of the HepPEd Program on HCV testing and treatment uptake amongst people incarcerated in Australian prisons, as well as changes in knowledge, attitudes, and capabilities of healthcare providers, correctional officers, and people in prison. The study is a controlled before and after study being conducted in 3-6 correctional centres in Australia.

DETAILED DESCRIPTION:
The National Prisons Hepatitis Education Program (HepPEd Program) is a national, prison-based hepatitis C health literacy education program for healthcare providers, correctional officers, and people in prison.

The broad goal of HepPEd: Research Evaluation is to measure the impact of a prison-specific hepatitis C (HCV) education program (the HepPEd Program) on enhancing HCV testing and treatment rates in Australian prisons. The HepPEd Program aims to improve HCV testing and treatment rates by enhancing the public health literacy of the prison sector regarding HCV in the prisons (that is the knowledge, attitudes and behaviours), and specifically targets the three key audience groups from the prison setting: healthcare providers, correctional officers, and people in prison.

The study will be conducted as a prison-level, controlled before-and-after trial with a primary objective of evaluating the impact of the HepPEd Program on HCV treatment uptake amongst people incarcerated in Australian prisons. Three to six Australian correctional centres will be selected to participate in the 9-month study. Each correctional centre will have a 3-month period of pre-intervention surveillance, involving monthly observation of HCV treatment uptake under existing operations. This will be followed by a three-month period of education delivery of the HepPEd Program (the 'education intervention'). The monthly surveillance data collection will continue during the intervention period. Finally, each correctional centre will have another 3-month period of post-intervention surveillance, again involving monthly surveillance of HCV treatment rates. Surveys will be conducted with members from each target audience group before and after the education intervention and dried blood spot testing will be conducted with members from the people in prison group to assess baseline HCV prevalence before the education intervention.

ELIGIBILITY:
All healthcare providers, correctional officers, and people in prison at the participating prison sites are anticipated to be exposed to the various HepPEd Program resources during the 3 month education intervention phase.

Participating prison sites must meet the following inclusion criteria to be eligible to participate in the study. Participating prison sites must have:

* a prisoner population of 400-600 inmates (assumed mean 500); and
* an existing prison-based hepatitis service undertaking both HCV testing and treatment.

Prisoners must meet the following inclusion criteria to be eligible to participate as peer educators. Prisoners must:

* be currently incarcerated in a participating correctional centre;
* anticipate being in the participating correctional centre for >12 months;
* be considered as capable and willing, and well-respected amongst their peers; and
* have approval from custodial authorities to participate as a peer educator.

Correctional officers must meet the following inclusion criteria to be eligible to participate as peer champions. Correctional officers must:

* be currently working in a participating correctional centre; and
* be considered as capable and willing, and well-respected amongst their peers.

Prisoners must meet the following inclusion criteria to be eligible to participate in the interview-style survey and dried blood spot (DBS) testing component:

1. be over the age of 18 years;
2. be currently incarcerated in a participating correctional centre;
3. have sufficient English comprehension skills to understand the survey questions; and
4. be willing and able to provide written informed consent.

Healthcare providers and correctional officers must meet the following inclusion criteria to be eligible to participate in the survey component:

1) be currently working in a participating correctional centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The change in the proportion of prisoners treated for HCV before and after the education intervention. | 9 months from baseline
  This will be measured by calculating the change in HCV treatment rates before and after the education intervention.

SECONDARY OUTCOMES:
The proportion of prisoners tested for HCV before and after the education intervention. | 9 months from baseline
  This will be measured by calculating the change in HCV testing rates before and after the education intervention.
The health literacy (knowledge, attitudes, and capabilities) amongst target audience groups (healthcare providers, correctional officers, and people in prison) before and after the education intervention. | 9 months from baseline
  This will be measured by assessing the change in health literacy before and after the education intervention.
The acceptability, utility, and impact of the HepPEd Program. | 9 months from baseline
  This is measured by surveys, before and after the education intervention.
The dose, reach, and fidelity of the HepPEd Program. | 9 months from baseline
  This is measured by surveys, before and after the education intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Capricornia Correctional Centre, Rockhampton, Queensland
  - Risdon Prison Complex, Hobart, Tasmania

IPD SHARING:
Plan to Share IPD: No